CLINICAL TRIAL: NCT02905188
Title: Glypican 3-specific Chimeric Antigen Receptor Expressing T Cells As Immunotherapy for Patients with Hepatocellular Carcinoma
Brief Title: Glypican 3-specific Chimeric Antigen Receptor Expressing T Cells for Hepatocellular Carcinoma (GLYCAR)
Acronym: GLYCAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Tannaz Armaghnay, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-38942 GLYCAR
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; GPC3-CAR T cells; GPC3-positive hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GLYCAR T cells + Fludarabine and Cytoxan (Experimental): GPC3-CAR (GLYCAR T cells) along with lymphodepleting chemotherapy (Cytoxan and Fludarabine) will be administered to patients with hepatocellular carcinoma.
  Interventions: Genetic: GLYCAR T cells; Drug: Cytoxan; Drug: Fludarabine

INTERVENTIONS:
Genetic: GLYCAR T cells — Five different dosing schedules will be evaluated. Three to six patients will be evaluated on each dosing schedule.
  The following dose levels will be evaluated:
  DL1: 1x10^7/m2
  DL2: 3x10^7/m2
  DL3: 1x10^8/m2
  DL4: 3x10^8/m2
  DL5: 1x10^9/m2
  If DLTs are observed on DL1, patients will be enrolled on DL0 at 3x10^6/m2 dose.
  The first patient on each dose level has to be 14 days post T-cell infusion before the second patient can be enrolled.
  The doses are calculated according to the actual number of GPC3-CAR transduced T cells.
  Other Names: GPC3-CAR T cells
Drug: Cytoxan — Cyclophosphamide will be given at a dose of 500 mg/m2/day for 3 days given intravenously
  Other Names: Cyclophosphamide
Drug: Fludarabine — Fludarabine will be given at a dose of 30 mg/m2/day for 3 days given intravenously

SUMMARY:
This study enrolls patients who have a type of cancer that arises from the liver called hepatocellular carcinoma. The cancer has come back, has not gone away after standard treatment, has spread outside of the liver or the patient cannot receive standard treatment. This research study uses special immune system cells called GLYCAR T cells, a new experimental treatment.

The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting cancer: antibodies and T cells. Antibodies are types of proteins that protect the body from infectious diseases and possibly cancer. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including cells infected with viruses and tumor cells. Both antibodies and T cells have been used to treat patients with cancers. They have shown promise, but have not been strong enough to cure most patients.

Investigators have found from previous research that they can put a new gene into T cells that will make them recognize cancer cells and kill them. In preclinical studies, the investigators made several genes called a chimeric antigen receptor (CAR), from an antibody called GC33 that recognizes glypican-3, a protein found on almost all hepatocellular carcinoma cells (GPC3-CAR). This study will test T cells genetically engineered with a GPC3-CAR (GLYCAR T cells) in patients with hepatocellular carcinoma.

The GLYCAR T cells are an investigational product not approved by the Food and Drug Administration.

The purpose of this study is to find the biggest dose of GLYCAR T cells that is safe, to see how long they last in the body, to learn what the side effects are and to see if the GLYCAR T cells will help people with GPC3-positive hepatocellular carcinoma.

DETAILED DESCRIPTION:
A maximum of 30 subjects will participate in the treatment part of this study.

Up to 180ml of blood is collected from patients to grow the T cells. The T cells are grown and a retrovirus (a special virus that can carry the GPC3 CAR gene into the T cells) is used to genetically engineer them. After the CAR gene is put into the T cells, the investigators make sure that they are able to kill hepatocellular carcinoma cells in the laboratory.

LYMPHODEPLETION CHEMOTHERAPY:

Several studies suggest that the infused T cells need room to be able to proliferate and accomplish their functions and that this may not happen if there are too many other T cells in circulation. Because of that, participants will receive treatment with cyclophosphamide (Cytoxan) and fludarabine for 3 days before receiving the T-cell infusion. These drugs will decrease the numbers of the participants' own T cells before the investigators infuse the GLYCAR T CELLS.

WHAT THE INFUSION WILL BE LIKE:

After making these cells, they will be frozen. If the patient agrees to participate in this study, at the time the patient is scheduled to be treated, the cells will then be thawed and injected into the patient over 1 to 10 minutes. The participant will receive the GLYCAR T CELLS 48-72 hours after completing the chemotherapy. The participant may be pretreated with Tylenol (acetaminophen) and Benadryl (diphenhydramine). Tylenol and Benadryl are given to prevent a possible allergic reaction to the T cell administration.

This is a dose escalation study, which means that the investigators do not know the highest dose of GLYCAR T cells that is safe. To find out, the investigators will give the cells to at least 3 participants at one dose level. If that is safe, they will raise the dose given to the next group of participants. The dose each patient gets will depend on how many participants get the agent before that patient and how they react. The investigator will tell each patient this information. This will help the patient think about possible harms and benefits. Since the treatment is experimental, what is likely to happen at any dose is not known.

All of the Treatments will be given by the Center for Cell and Gene Therapy at Houston Methodist Hospital.

Medical tests before treatment:

* Physical exam and History
* Blood tests to measure blood cells, kidney and liver function and blood clotting (INR).
* If the patient is infected with the hepatitis B virus (HBV) we will do a test to measure the levels of the virus
* Pregnancy test (if the patient is a female who can get pregnant)
* Measurements of the patient's tumor by scans (within 4 weeks before chemotherapy) and the tumor marker alfa-fetoprotein (AFP), if the patient's tumor produces this protein.
* Tumor biopsy

Medical tests during and after treatment:

* Physical exams and History
* Blood tests to measure blood cells, kidney and liver function and blood clotting (INR)
* If the patient is infected with the hepatitis B virus (HBV) we will do a test to measure the levels of the virus
* Measurements of the tumor maker alfa-fetoprotein (AFP), if the patient's tumor produces this protein
* Measurements of the patient's tumor by scans (8 weeks after the infusion +/- 1 week)
* Tumor biopsy (optional)

FOLLOW-UP STUDIES

The investigators will follow the participant during and after the injections. To learn more about the way the T cells are working in the participant's body, up to 60 mL (12 teaspoons) of blood will be taken from the participant before the chemotherapy, before the T-cell infusion, 3 to 4 hours after the infusion, 3 to 4 days after the infusion (this time point is optional ) at 1 week, 2 weeks, 4 weeks, 6 weeks and 8 weeks after the injection, every 3 months for 1 year, every 6 months for 4 years and then every year for the next 10 years. Total time participation for this study will be 15 years.

During the time points listed above, if the T cells are found in the participant's blood at a certain amount an extra 5mL of blood may need to be collected for additional testing.

The investigators will use this blood to look for the frequency and activity of the cells that they have given; that is, to learn more about the way the T cells are working and how long they last in the body. They will also use this blood to see if there are any long-term side effects of putting the new gene (chimeric antigen receptor, CAR) into the cells. In addition to the blood draws, because the participants have received cells that have had a new gene put in them, they will need to have long term follow up for 15 years so the investigators can see if there are any long term side effects of the gene transfer.

Once a year, participants will be asked to have their blood drawn and answer questions about their general health and medical condition. The investigators may ask participants to report any recent hospitalizations, new medications, or the development of conditions or illness that were not present when they enrolled in the study and may request that physical exams and/or laboratory tests be performed if necessary.

Prior to procurement we confirmed GPC3-expression in your tumor by obtaining part of a biopsy sample that was done for clinical purposes. We will obtain an additional tumor biopsy at 2 weeks after treatment for research purposes. These samples will be used to look for GPC3-CAR T cells in the tumor and to learn more about the effects of the treatment on your disease.

In the event that a tumor biopsy is performed for clinical reasons the investigators will request permission to obtain excess sample to learn more about the effects of the treatment on the participant's disease. In the event of death, the investigators will request permission to perform an autopsy to learn more about the effects of the treatment on the participant's disease and if there were any side effects from the cells with the new gene.

If participants develop a second abnormal cancer growth, significant blood or nervous system disorder during the trial, a biopsy sample of the tissue will be tested (if a sample can be obtained).

ELIGIBILITY:
Procurement Eligibility

Inclusion Criteria:

* Histology-proven hepatocellular carcinoma (HCC) which is unresectable, recurrent and/or metastatic
* Barcelona Clinic Liver Cancer Stage A, B or C
* GPC3-positive HCC
* Age ≥ 18 years
* Karnofsky score ≥ 60% (See appendix I)
* Life expectancy ≥ 12 weeks
* Child-Pugh-Turcotte score <8
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

Exclusion Criteria

* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment (only patients who have received prior therapy with murine antibodies).
* History of liver transplantation
* Known HIV positivity
* Active bacterial, fungal or viral infection (except Hepatitis B or Hepatitis C virus infections)
* Severe previous toxicity from cyclophosphamide or fludarabine

Treatment Eligibility

Inclusion Criteria:

* Histology-proven hepatocellular carcinoma (HCC) which is unresectable, recurrent and/or metastatic
* Barcelona Clinic Liver Cancer Stage A, B or C
* GPC3-positive HCC
* Age ≥ 18 years
* Life expectancy of ≥ 12 weeks
* Karnofsky score ≥ 60%
* Child-Pugh-Turcotte score < 8
* Adequate organ function:

  * creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 ml/min
  * serum AST< 5 times ULN
  * total bilirubin < 3 times ULN for age
  * INR ≤1.7
  * absolute neutrophil count > 500/microliter
  * platelet count > 20,000/microliter (can be transfused)
  * Hgb ≥7.0 g/dl (can be transfused)
  * Pulse oximetry >90% on room air
* Recovered from acute toxic effects of all prior antineoplastic drugs before entering this study (including investigational drugs) based on the enrolling physician's assessment (if some effects of chemotherapy are expected to last long term, patient is eligible if meeting other eligibility criteria).
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 3 months after the T-cell infusion.
* Available autologous transduced T cell product
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

Exclusion Criteria:

* Eligible for complete tumor resection or liver transplantation.
* Pregnancy or lactation (for women at child-bearing age, birth control is required)
* Hepatic encephalopathy
* Uncontrolled infection
* Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day)
* Known HIV positivity
* Active bacterial, fungal or viral infection (except Hepatitis B or Hepatitis C virus infections)
* History of liver transplantation
* Heart failure of Class III-IV and / or C-D per NYHA Criteria
* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment (only patients who have received prior therapy with murine antibodies)
* Severe previous toxicity from cyclophosphamide or fludarabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | 6 weeks
  DLT will be defined as any of the following that may, after consultation with the FDA, be considered possibly, probably, or definitely related to the study cellular products.
  * Any Grade 5 event
  * Non-hematologic dose-limiting toxicity is any Grade 3 or Grade 4 non-hematologic toxicity that fails to return to Grade 2 within 72 hours
  * Grade 2 to 4 allergic reaction to CAR T cell infusion.
  * Hematologic dose limiting toxicity is defined as any Grade 4 hematologic toxicity that fails to return to Grade 2 or baseline (whichever is more severe) within 14 days.
  * Grade 3 and 4 expected reactions due to CRS and neurotoxicity are seen with the use of CAR-based immunotherapy. Grade 3 cytokine release syndrome (CRS) infusion reactions and neurologic toxicity will only be reported to the FDA if they fail to return to Grade 1 within 7 days. Grade 4 CRS and neurologic toxicities will be reported to the FDA in an expedited fashion.
Recommended Phase 2 Dose (RP2D) | 2 years
  The RP2D is based upon the review of all available data including safety, preliminary anti-tumor activity, and MTD.

SECONDARY OUTCOMES:
Percent of Patients with best response as either complete remission or partial remission | 6 weeks
  Response rates will be estimated as the percent of patients whose best response is either complete remission or partial remission by combining the data from the two patients. To compare with historical data, a 95% confidence interval will be calculated for the response rate.
Median T cell persistence | 15 years
  as measured by PCR

CONTACTS AND LOCATIONS:
Overall Officials: Tannaz Armaghany, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No